CLINICAL TRIAL: NCT03169608
Title: Predicting Post-surgery Complications in Patients Undergoing Coronary Artery Bypass Graft Through the Assessment of Perioperative Cardiovascular Control Indices
Brief Title: Autonomic State, Cardiovascular Control and Outcomes in Coronary Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director of Cardiothoracic Anesthesia and ICU Dept, IRCCS Policlinico S. Donato
Other Study IDs: GR2013; GR-2013-02356272 (Other Grant/Funding Number: Italian Ministery of Health)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Atrial Fibrillation; Acute Kidney Injury
Keywords: autonomic nervous system; atrial fibrillation; acute kidney injury; baroreflex sensitivity; microcirculation; coronary artery bypass graft
MeSH Terms: conditions — Atrial Fibrillation; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Characterization of the perioperative autonomic nervous system state, cardiovascular and cerebrovascular control and microcirculation in order to predict postoperative atrial fibrillation and acute kidney injury in patients undergoing coronary artery bypass graft surgery

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and acute kidney injury (AKI) are common postoperative complications in patients undergoing coronary artery bypass graft (CABG) surgery. AKI increases postoperative mortality and AF prolongs the hospital stay.

Autonomic dysfunction, baroreflex impairment and an inadequate microvascular perfusion may play a relevant role in triggering AF and AKI.

The perioperative characterization of the autonomic nervous system (ANS) and of the microcirculation might improve risk stratification and help in the prevention and early treatment of AF and AKI in CABG surgery.

The study aims are: i) to collect a number of perioperative indices describing the state of the ANS and of the microcirculation; ii) to assess the correlation among the different indices and their association with AF and AKI; iii) to develop a predictive model of postoperative outcomes (AF and AKI) accounting for perioperative autonomic indices and microcirculatory variables.

Population: 200 adults subjects scheduled for CABG surgery, with or without additional intervention Methods: perioperative (in the operating room) acquisition of ECG, arterial blood pressure, cerebral blood flow velocity as derived from transcranial doppler technique, microcirculation parameters as derived from sidestream dark field images Statistics: receiver operating characteristic (ROC) curve analysis with adequate cut-off values

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* sinus rhythm
* absence of pathologies affecting autonomic nervous system (e.g. diabetes with neuropathy)
* informed consent signed
* elective or urgent surgery

Exclusion Criteria:

* age under 18
* absence of sinus rhythm
* pathologies affecting autonomic nervous system
* emergency surgery (to be operated immediately)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult coronary surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-07-14 (Estimated); Study Completion 2019-07-14 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation | from the admission to the ICU to the hospital discharge, with an average of 8 days
  any atrial fibrillation event recorded during the postoperative period, as derived from ECG monitoring
Acute Kidney Injury | 48 hours from surgery
  50% increase of serum creatinine with respect to baseline or absolute increase > 0.3 mg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, FESC, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villareal RP, Hariharan R, Liu BC, Kar B, Lee VV, Elayda M, Lopez JA, Rasekh A, Wilson JM, Massumi A. Postoperative atrial fibrillation and mortality after coronary artery bypass surgery. J Am Coll Cardiol. 2004 Mar 3;43(5):742-8. doi: 10.1016/j.jacc.2003.11.023. PMID 14998610
- [Background] Provenchere S, Plantefeve G, Hufnagel G, Vicaut E, de Vaumas C, Lecharny JB, Depoix JP, Vrtovsnik F, Desmonts JM, Philip I. Renal dysfunction after cardiac surgery with normothermic cardiopulmonary bypass: incidence, risk factors, and effect on clinical outcome. Anesth Analg. 2003 May;96(5):1258-1264. doi: 10.1213/01.ANE.0000055803.92191.69. PMID 12707117
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Pagani M, Montano N, Porta A, Malliani A, Abboud FM, Birkett C, Somers VK. Relationship between spectral components of cardiovascular variabilities and direct measures of muscle sympathetic nerve activity in humans. Circulation. 1997 Mar 18;95(6):1441-8. doi: 10.1161/01.cir.95.6.1441. PMID 9118511
- [Background] Faes L, Porta A, Rossato G, Adami A, Tonon D, Corica A, Nollo G. Investigating the mechanisms of cardiovascular and cerebrovascular regulation in orthostatic syncope through an information decomposition strategy. Auton Neurosci. 2013 Nov;178(1-2):76-82. doi: 10.1016/j.autneu.2013.02.013. Epub 2013 Mar 27. PMID 23541295
- [Background] Ince C. The microcirculation is the motor of sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S13-9. doi: 10.1186/cc3753. Epub 2005 Aug 25. PMID 16168069
- [Derived] Singh P, Porta A, Ranucci M, Cairo B, Gelpi F, Caruso R, Magon A, Baroni I, Conte G, Bari V. Identifying and preliminary validating patient clusters in coronary artery bypass grafting: integrating autonomic function with clinical and demographic data for personalized care. Eur J Cardiovasc Nurs. 2025 Sep 5;24(6):898-910. doi: 10.1093/eurjcn/zvaf059. PMID 40186491